CLINICAL TRIAL: NCT03147378
Title: Food-effect Study of Weekly Administration of (bi-)Daily Oral Docetaxel (ModraDoc006) in Combination With Ritonavir
Brief Title: Food Effect Study of ModraDoc006 in Combination With Ritonavir
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Modra Pharmaceuticals (Industry)
Collaborators: The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: N15FED
Record Dates: First submitted 2017-05-02; First posted 2017-05-10 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Solid Tumor, Adult

STUDY DESIGN:
Intervention Model Description: After randomization eight patients will receive ModraDoc006/r in fasting condition week 1 and in fed condition week 2, and another eight patients will receive ModraDoc006/r in fed condition week 1 and in fasting condition week 2
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- arm A Fasting-Fed condition (Experimental): ModraDoc006/r will be administered in fasting condition week 1 and in fed condition week 2
  Interventions: Drug: ModraDoc006/r
- arm B Fed-Fasting condition (Experimental): ModraDoc006/r will be administered in fed condition week 1 and in fasting condition week 2
  Interventions: Drug: ModraDoc006/r

INTERVENTIONS:
Drug: ModraDoc006/r — Treatment with weekly ModraDoc006 (oral docetaxel) 10mg tablets in combination with ritonavir 100mg tablets in fed or fasting condition
  Other Names: oral docetaxel formulation

SUMMARY:
This study aims to evaluate the effect of food on the pharmacokinetics of ModraDoc006 in combination with ritonavir, in an open-label, cross-over design. Patients will be randomized into two treatment groups receiving ModraDoc006/r week 1 under fasting and week 2 under fed condition, or vice versa.

DETAILED DESCRIPTION:
In this study the effect of food on the plasma exposure of ModraDoc006/ritonavir will be assessed in an open-label, cross-over design. Patients will receive ModraDoc006/ritonavir at the dose of 30 mg ModraDoc006 with 100 mg ritonavir.

Patients will be randomized 1:1 into two treatment groups (in total 16 evaluable patients are needed):

* Group A: will receive ModraDoc006/ritonavir under fasting conditions the first week and in a fed condition the second week of treatment.
* Group B: will receive ModraDoc006/ritonavir under fed condition the first week and under fasted condition the second week of treatment.

The department of pharmacy of The Netherlands Cancer Institute - Antoni van Leeuwenhoek Hospital has developed a solid oral dosage form of docetaxel, ModraDoc006 10 mg tablets. This formulation has been investigated in two phase I clinical studies in combination with the CYP3A4 inhibitor ritonavir, according to a weekly once-daily (QD) or bi-daily (BID) schedule, respectively. Maximum Tolerated Dose (MTD) and pharmacokinetics of both regimes have been determined and further clinical testing is being planned, in particular of the weekly bi-daily regime.

The aim of the current study is to evaluate the effect of food on the pharmacokinetics of ModraDoc006 in combination with ritonavir. For the ritonavir tablet formulation used in this trial a food-effect on the bio-availability has been found in two prior studies. In these trials the plasma concentrations were lower when ritonavir was given after a moderate or high-fat meal. Plasma concentrations and T-lag were dependent on the type/amount of food administered. Concentrations were lower and T-lag longer when a high-fat meal was administered as compared to a moderate fat meal.

Randomization will be performed centrally at the Biometrics Department of the Netherlands Cancer Institute using a minimization technique as implemented in TENALEA©.

Pharmacokinetics will be performed in week 1 and 2 for up to 48 hours after study drug administration (see Pharmacokinetics paragraph for exact time points). Patients will receive a high-fat meal on the morning of the day of fed condition pharmacokinetics, half an hour prior to intake of ModraDoc006/ritonavir.

After week 2, the N15FED study will be completed and patients can be enrolled in the roll over study N17DEX to continue their treatment with ModraDoc006/r (at the dose of BID 30/20 mg ModraDoc006 in combination with BID 100 mg ritonavir) in their best interest and to assess the long-term safety of this treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Histological or cytological proof of cancer
2. Patients for whom no standard therapy of proven benefit exists
3. Patients who might benefit from treatment with docetaxel, e.g. advanced breast, gastric, esophagus, bladder, ovarian cancer and non-small cell lung cancer, head and neck cancers, prostate cancer and carcinoma of unknown primary site.
4. Age 18 years
5. Able and willing to give written informed consent
6. Able and willing to undergo blood sampling for pharmacokinetics
7. Life expectancy 3 months
8. Minimal acceptable safety laboratory values 8.1. Hb ≥ 6.0 mmol/l 8.2. ANC 1.5 x 109 /L 8.3. Platelet count 100 x 109 /L 8.4. Serum bilirubin 1.5 x ULN, ALAT and ASAT 2.5 x ULN (or 5 x ULN in case of presence of liver metastases) 8.5. Serum creatinine 1.5 x ULN or creatinine clearance 50 ml/min (by Cockcroft-Gault formula).
9. WHO performance status of 1
10. No radio- or chemotherapy within the last 4 weeks prior to first dose of study medication (palliative radiation on limited field for pain reduction is allowed)
11. Able and willing to swallow oral medication.

Exclusion Criteria:

1. Patients with known alcoholism, drug addiction and/or psychotic disorders in the medical history that are not suitable for adequate follow up
2. Women who are pregnant or breast-feeding.
3. Men and women, who do not agree to use two reliable contraceptive methods hroughout the study (adequate contraceptive methods are: use of oral, injected or implanted hormonal methods of contraception, placement of an intrauterine device (IUD) or intrauterine system (IUS), barrier methods of contraception: condom, diaphragm with spermicide, male sterilization, true abstinence).
4. Concomitant use of MDR and CYP3A modulating drugs such as Ca+-entry blockers (verapamil, dihydropyridines), cyclosporine, quinidine, quinine, tamoxifen, megestrol and grapefruit juice, concomitant use of HIV medications; other protease inhibitors, (non) nucleoside analogs, St. Johns wort or macrolide antibiotics like erythromycin and clarithromycin.
5. Uncontrolled infectious disease or known HIV-1 or HIV-2 infection
6. Unresolved (>grade 1) toxicities of previous chemotherapy, excluding alopecia
7. Bowel obstructions or motility disorders or previous surgery that may influence the absorption of drugs
8. Neurologic disease that may render a patient at increased risk for peripheral or central neurotoxicity
9. Pre-existing neuropathy greater than CTC grade 1
10. Patients with suspected or known brain metastases, unless they have been adequately treated and are asymptomatic without use of corticosteroids (for at least 1 month)
11. Evidence of any other disease, neurological or metabolic dysfunction, physical examination finding or laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or puts the patient at high risk for treatment-related complications.
12. Legal incapacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-05-10 (Actual); Primary Completion 2018-04-04 (Actual); Study Completion 2018-04-04 (Actual)

PRIMARY OUTCOMES:
The AUC of docetaxel (area under the curve) | Pharmacokinetic sampling during 2 weeks, 0-48 hours after administration (i.e. the 2 treatment cycles)
  The AUC of docetaxel given as bi-daily ModraDoc006 10 mg tablets in combination with ritonavir after administration in a high fed and fasting condition
The cMax (peak concentration) of docetaxel | Pharmacokinetic sampling during 2 weeks, 0-48 hours after administration (i.e. the 2 treatment cycles)
  The cMax (peak concentration) of docetaxel given as bi-daily ModraDoc006 10 mg tablets in combination with ritonavir after administration in a high fed and fasting condition

SECONDARY OUTCOMES:
The hematological and non-hematological toxicity profile of oral docetaxel in combination with ritonavir | Safety and tolerance will be evaluated during the complete study treatment untill 28 days after the last intake, using the CTCAEv4.03 grading system
  The number of CTCAE v.4.03 grade 3-4 toxicities during treatment with ModraDoc006/r
The effect of functional genetic polymorphisms on the pharmacokinetics of oral docetaxel and ritonavir (to understand the mechanism of the drug-drug interaction more thoroughly) | Sampling at baseline, the analyses will be performed retrospectively
  Pharmacogenetic analyses will be performed for polymorphisms in drug metabolizing enzymes (e.g., but not limited to genes encoding for P-glycoprotein (ABCB1/MDR1), Multidrug resistance protein 2 (ABCC2/MRP2), Organic anion-transporting polypeptides 1B3 (OATP1B3), Cytochrome P450 (CYP) 3A4 and CYP3A5)

CONTACTS AND LOCATIONS:
Overall Officials: Serena Marchetti, MD, PhD, Principal Investigator — The Netherlands Cancer Institute
Locations (1):
- Netherlands Cancer Institute - Antoni van Leeuwenhoek, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vermunt MAC, de Weger VA, Janssen JM, Lopez-Yurda MI, Keessen M, Thijssen B, Rosing H, Huitema ADR, Beijnen JH, Marchetti S. Effect of Food on the Pharmacokinetics of the Oral Docetaxel Tablet Formulation ModraDoc006 Combined with Ritonavir (ModraDoc006/r) in Patients with Advanced Solid Tumours. Drugs R D. 2021 Mar;21(1):103-111. doi: 10.1007/s40268-020-00336-x. Epub 2021 Jan 19. PMID 33464545